CLINICAL TRIAL: NCT00361361
Title: The Efficacy of 308nm Excimer Laser in White Striae
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr.Nima Ostovari
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: src-ost-1360
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2006-11

CONDITIONS: White Striae; Excimer Laser

INTERVENTIONS:
Device: Excimer Laser Therapy — excimer laser is a UV 308nm laser. repeated sessions (10 sessions) needed. once per week.

SUMMARY:
The purpose of this study is to determine whether 308nm Excimer Laser therapy are effective in the color correction of white striae.

DETAILED DESCRIPTION:
The use of excimer laser in modified program in white striae during a few months.

ELIGIBILITY:
Inclusion Criteria:

* White Striae

Exclusion Criteria:

* Red Striae

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-07; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Clinical darkening of striaes

SECONDARY OUTCOMES:
Colorimetric assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nima Ostovari, M.D., Study Director — Shahid Beheshti University of Medical Sciences; Parviz Toossi, MD, Study Chair — skin research center of shaheed-beheshti medical university
Locations (1):
- Skin Research Center, Shaheed Beheshti Medical University, Tehran, Iran